CLINICAL TRIAL: NCT03629808
Title: The Effect of Residual Gastric Antrum Size During Laparoscopic Sleeve Gastrectomy in Reducing Postoperative Gastrointestinal Symptoms: a Cohort Study
Brief Title: Laparoscopic Sleeve Gastrectomy: a Cohort Study
Status: Completed | Type: Observational
Sponsor: Beijing Friendship Hospital (Other)
Collaborators: Peking Union Medical College Hospital (Other); Beijing Tiantan Hospital (Other); Beijing Hospital (Other Government); Beijing Shijitan Hospital, Capital Medical University (Other)
Responsible Party: Principal Investigator, Zhongtao Zhang, Director of general surgery, principal investigator, Beijing Friendship Hospital
Other Study IDs: BFH-LSG 01
Record Dates: First submitted 2018-07-17; First posted 2018-08-14 (Actual); Last update posted 2020-04-22 (Actual); Status verified 2020-04

CONDITIONS: Laparoscopic Sleeve Gastrectomy
Keywords: metabolic surgery; laparoscopic sleeve gastrectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group1: 4-6cm: 4-6cm from starting point of gastrectomy to pylorus
  Interventions: Procedure: 4-6cm from starting point of gastrectomy to pylorus
- Group2: 2-4cm: 2-4cm from starting point of gastrectomy to pylorus
  Interventions: Procedure: 2-4cm from starting point of gastrectomy to pylorus

INTERVENTIONS:
Procedure: 4-6cm from starting point of gastrectomy to pylorus — The starting point of gastrectomy of the distance from the pylorus is 4-6cm during operative.
  Groups: Group1: 4-6cm
Procedure: 2-4cm from starting point of gastrectomy to pylorus — The starting point of gastrectomy of the distance from the pylorus is 2-4cm during operative.
  Groups: Group2: 2-4cm

SUMMARY:
This is a prospective cohort study, which subjects were obese patients requiring LSG surgery. LSG with different gastric resection starting points (2-4cm/4-6 cm from pylorus) as intervention method. The main observation is the incidence and extent of upper gastrointestinal symptoms (such as nausea, vomiting, retching, reflux, difficulty swallowing, etc.).In addition, secondary observations include the excess weight loss (%EWL) and postoperative complications. Aim to investigate the effects of LSG surgery in different starting points of gastric resection on postoperative upper gastrointestinal symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Patients were accepted for surgery if they satisfied the guidelines of the Society of Chinese Gastroenterological Surgeons [body mass index (BMI) ≥40 kg/m2 or BMI ≥35 kg/m2 with at least one co-morbidity associated with obesity (type 2 diabetes, hypertension, dyslipidemia, obstructive sleep apnea), age between 18 and 60 years, and failure of conservative treatment over 2 years].
* All patients undergo preoperative upper gastrointestinal (GI) endoscopy.

Exclusion Criteria:

* any patient who had previously been submitted to any type of bariatric surgery;
* patient currently taking anti-nausea or GERD medications preoperatively;
* any current smokers；
* active duodenal/gastric ulcer disease；
* difficult to treat gastroesophageal reflux disease (GERD) with a large hiatal hernia；
* previous major gastrointestinal surgery；
* diagnosed or suspected malignancy；
* poorly controlled significant medical or psychiatric disorders；
* disorders such as a medical history of major pathology;
* can not be able to understand and willing to participate in this registry with signature.

Ages: 15 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population will comprise male and non-pregnant female patients, aged 16-65years both inclusive, with morbid obesity.
Sampling Method: Non-Probability Sample
Enrollment: 138 (Actual)
Dates: Start 2018-07-10 (Actual); Primary Completion 2020-03-28 (Actual); Study Completion 2020-04-20 (Actual)

PRIMARY OUTCOMES:
The incidence rate of upper gastrointestinal symptoms after surgery | 1 year after surgery
  We use three scales to evaluate the incidence of upper gastrointestinal symptoms,include the Chinese translation of R-INVR(the Index of Nausea, Vomiting, and Retching)、EAT-10(Validity and Reliability of the Eating Assessment Tool) and GIS(GERD impact serve).These three scales describe postoperative upper gastrointestinal symptoms,which include vomiting, dysphagia,and acid reflux,heartburn.We focus on the incidence rate of the above symptoms in one year after surgery during 1 year.
  Visit: Post-op 12 months Visit(±7 Days)

SECONDARY OUTCOMES:
The excess weight loss (%EWL) after surgery | 1 year after surgery
  Percent excess weight loss (%EWL), %EWL=[(initial weight)-(post-op weight)]/[(initial weight)-(ideal weight)] (in which "ideal weight" is defined by the weight corresponding to a BMI of 25 kg/m2).
  Visit 1: Baseline Visit (Day 0-1) Visit 2: Post-op 3 days Visit Visit 3: Post-op 7 days Visit Visit 4: Post-op 1 month Visit(±3 Days) Visit 5: Post-op 3 months Visit(±7 Days) Visit 6: Post-op 12 months Visit(±7 Days)
the rate of postoperative complications after surgery | 1 year after surgery
  Postoperative complications including but not limited to: 1, abdominal bleeding; 2, gastrointestinal bleeding; 3, intestinal obstruction; 4, digestive tract leakage 5, anastomotic stenosis / gastric stenosis; 6, death ,etc.
  Visit 1: Baseline Visit (Day 0-1) Visit 2: Post-op 3 days Visit Visit 3: Post-op 7 days Visit Visit 4: Post-op 1 month Visit(±3 Days) Visit 5: Post-op 3 months Visit(±7 Days) Visit 6: Post-op 12 months Visit(±7 Days)
The extent of upper gastrointestinal symptoms after surgery | 1 year after surgery
  We use three scales to evaluate the incidence of upper gastrointestinal symptoms,include the Chinese translation of R-INVR(the Index of Nausea, Vomiting, and Retching)、EAT-10(Validity and Reliability of the Eating Assessment Tool) and GIS(GERD impact serve).These three scales quantify the degree of vomiting, difficulty swallowing, acid reflux, heartburn, etc.We will calculate the extent of the above upper gastrointestinal symptoms at five time points in one year after surgery.
  Visit 1: Post-op 3 days Visit Visit 2: Post-op 7 days Visit Visit 3: Post-op 1 month Visit(±3 Days) Visit 4: Post-op 3 months Visit(±7 Days) Visit 5: Post-op 12 months Visit(±7 Days)

CONTACTS AND LOCATIONS:
Overall Officials: Zhongtao Zhang, Principal Investigator — Beijing Friendship Hospital
Locations (1):
- Beijing Friendship Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Result] Chow, S.C.; Shao, J.; Wang, H. 2003. Sample Size Calculations in Clinical Research. Marcel Dekker. New York.